CLINICAL TRIAL: NCT07018999
Title: Immersive Virtual Reality Exposure for Reducing Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Collaborators: The Hong Kong Polytechnic University (Other); City University of Hong Kong (Other)
Responsible Party: Principal Investigator, KWOK, Vansie, Consultant, Hong Kong Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HKCH-REC-2021-026; KCC/RC/G/2223-B05 (Other Grant/Funding Number: Hospital Authority Kowloon Central Cluster Research Grant)
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety State; Satisfaction; Compliance
Keywords: Virtual reality; perioperative anxiety; children
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to intervention group (VR group) and conventional group (Non-VR group). Participants assigned to the VR group will watch the designed VR immersive experience with headset, whereas participants assigned to the non-VR group will receive standard medical care without any additional intervention.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) group (Experimental): Participants assigned to the VR group will watch the designed VR immersive experience with headset on the day of surgery on top of the usual interventions as received in the control group.
  Interventions: Device: Immersive virtual reality operating theatre tour
- Control group (No Intervention): All recruited participants will receive standard medical care and provided with information regarding the perioperative journey as per usual practice, including watching an introductory video in the waiting room area with accompanying adults, receiving perioperative education by a pre-anaesthetic nurse, as well as having an opportunity to have any questions answered by an anaesthesiologist in the pre-anaesthetic assessment clinic. They will not receive Virtual Reality intervention before surgery on surgery day

INTERVENTIONS:
Device: Immersive virtual reality operating theatre tour — In a joint project involving the Department of Computing of Hong Kong Polytechnic University, the Department of Computer science Center for Innovative Applications of Internet and Multimedia Technologies of the City University of Hong Kong and the Hong Kong Children's Hospital (HKCH), an immersive VR operating theatre tour will be designed as part of preoperative education for participants. A simulation of the perioperative journey in HKCH operating theatre will be created to help participants form realistic expectations of their perioperative journey, and virtual exposure of different medical equipment helps participants cope with their worries for the anticipated procedures. Parents/legal guardians will be able to monitor the VR experience on tablets via the monitoring software, which displays what the participants see in VR.
  Arms: Virtual reality (VR) group

SUMMARY:
Perioperative anxiety management for children undergoing surgery poses a major challenge to anaesthesiologists as high anxiety, reported in numerous studies, leads to detrimental effects physiologically, mentally and on pain scores. Traditional methods, including administration of anxiolytics pre-op has its own limitations e.g. side effects of drugs. Non-pharmacological approaches e.g. OT orientation or information have a heavy reliance on manpower. A sustainable and reliable non-pharmacological method that requires minimal manpower support is needed for the effective management of paediatric perioperative anxiety.

Virtual reality utilises a head-mounted display with visual, auditory and tactile stimuli to simulate a fully immersive 3-dimensional environment. Its application in the paediatric perioperative setting can be either as a distraction during painful procedures or during induction of anaesthesia or as an exposure tool in preoperative education and has demonstrated success in literature.

In a joint project involving the Department of Computing of Hong Kong Polytechnic University, the Department of Computer Science Center for Innovative Applications of Internet and Multimedia Technologies of the City University of Hong Kong and the Hong Kong Children's Hospital (HKCH), an immersive VR operating theatre tour will be designed as part of preoperative education for children. A simulation of the perioperative journey in HKCH operating theatre will be created to help children form realistic expectations of their perioperative journey to cope with their worries about the anticipated procedures.

DETAILED DESCRIPTION:
Undergoing an operation is a major stress for both children and their families, with up to 50% of the children reported to have significant perioperative anxiety . High levels of perioperative anxiety in children manifest as tension, irritability and increased autonomic nervous system activity; and are associated with a multitude of adverse clinical outcomes, including increased postoperative analgesia requirement, increased postoperative emergence delirium, increased postoperative behavioural changes (e.g. nightmares, postoperative separation and general anxiety, eating problems that can persist up to 2 weeks after surgery). Furthermore, it impacts patient and parental satisfaction, creating an overall negative experience for families and staff.

The multifaceted risk factors of perioperative anxiety in children warrant a multi-modal array of tools up anaesthesiologists' sleeves to tailor for different children's needs based on age, understanding of instructions, and temperament . While pharmacological anxiolytics, e.g. Dexmedetomidine and Midazolam, are commonly deployed and effective, it has its limitations, such as time to effect, patient's age, as well as paradoxical agitation reported up to 10% for Midazolam, as well as taking away a learning opportunity for children to cope with stress. Common non-pharmacological approaches include parental presence during induction of anaesthesia, distraction techniques, and educational approaches.

Traditional educational approaches often involve providing information to children and parents/legal guardians by written pamphlets, either physical or video tour of the operating room, recovery area, and orientation of medical equipment. With the advance of technology, children are often familiar and easily engaged with technological devices, including smart phones, tablets, video games, and even immersive virtual reality (VR). VR is increasingly utilized in clinical setting, providing a fun and engaging educational experience for children.

VR utilizes a head-mounted display with visual, auditory and tactile stimuli to simulate a fully immersive 3-dimensional environment. Its application in the paediatric perioperative setting can be either as distraction during painful procedures or during induction of anaesthesia, or as an exposure tool in preoperative education. A meta-analysis of the effect of VR on preoperative anxiety shows a significant reduction of preoperative anxiety in paediatric patients. Previous study utilized a famous cartoon character in the VR preoperative educational video and showed significant reduction in preoperative anxiety when compared to children receiving information through conventional means. This benefit of VR exposure in reducing preoperative anxiety is not only evident in numerous studies measuring anxiety score, but also demonstrated in studies measuring salivary cortisol concentration.

In a joint project involving the Department of Computing of Hong Kong Polytechnic University, the Department of Computer science Center for Innovative Applications of Internet and Multimedia Technologies of the City University of Hong Kong and the Hong Kong Children's Hospital (HKCH), an immersive VR operating theatre tour will be designed as part of preoperative education for children. A simulation of the perioperative journey in HKCH operating theatre will be created to help children form realistic expectations of their perioperative journey, and virtual exposure of different medical equipment helps children cope with their worries for the anticipated procedures. Parents/legal guardians will be able to monitor the VR experience on tablets via the monitoring software, which displays what the children see in VR. Given the fact that the capacity of conventional approaches, e.g. child-play involvement by child-life specialists are hugely limited now due to COVID pandemic, such a VR-enabled approach may help to alleviate patient's anxiety.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologist (ASA) physical status I or II
* Undergo elective surgical procedures which requires general anaesthesia
* No previous experience of anaesthesia or surgery

Exclusion Criteria:

* Patients who are undergoing ultra-major surgery requiring postoperative intensive care unit care.
* Patients who are blind, or with hearing impairment
* Patients with significant developmental or cognitive delays, ADHD or autism
* Patients with history or current symptoms of vertigo
* Patients with history of epilepsy or seizures
* Patients who require anxiolytic premedication
* Patients who have physical conditions that prohibit use of headsets e.g. head / facial injuries, open skin or infectious condition on head/face, head/ facial malformation that precludes proper fitting of the VR headset
* Non-Cantonese speaking patients (due to limited resources of having Cantonese speaking VR design)
* Patients and/or parents/legal guardians who refuse to participate in study

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vansie Kwok, MBBS, FHKCA, Principal Investigator — Department of Anaesthesiology & Perioperative Medicine, Hong Kong Children's Hospital; Richard C Li, MSc, PhD, Principal Investigator — Department of Computing, Hong Kong Polytechnic University
Locations (1):
- Operating Theatre, Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in final publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1-2 Years of Trial Completion
Access Criteria: Interested individual will be able to access the IPD by direct e-mail contact with principal investigators.

REFERENCES:
- [Background] Moura LA, Dias IM, Pereira LV. Prevalence and factors associated with preoperative anxiety in children aged 5-12 years. Rev Lat Am Enfermagem. 2016 Jun 14;24:e2708. doi: 10.1590/1518-8345.0723.2708. PMID 27305179
- [Background] Kain ZN, Mayes LC, Wang SM, Caramico LA, Hofstadter MB. Parental presence during induction of anesthesia versus sedative premedication: which intervention is more effective? Anesthesiology. 1998 Nov;89(5):1147-56; discussion 9A-10A. doi: 10.1097/00000542-199811000-00015. PMID 9822003
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Yuan JC, Rodriguez S, Caruso TJ. Unique considerations of virtual reality utilization for perioperative pediatric patients. Paediatr Anaesth. 2021 Mar;31(3):377-378. doi: 10.1111/pan.14108. No abstract available. PMID 33631038
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Ganry L, Hersant B, Sidahmed-Mezi M, Dhonneur G, Meningaud JP. Using virtual reality to control preoperative anxiety in ambulatory surgery patients: A pilot study in maxillofacial and plastic surgery. J Stomatol Oral Maxillofac Surg. 2018 Sep;119(4):257-261. doi: 10.1016/j.jormas.2017.12.010. Epub 2018 Jan 6. PMID 29317347
- [Background] Eijlers R, Dierckx B, Staals LM, Berghmans JM, van der Schroeff MP, Strabbing EM, Wijnen RMH, Hillegers MHJ, Legerstee JS, Utens EMWJ. Virtual reality exposure before elective day care surgery to reduce anxiety and pain in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):728-737. doi: 10.1097/EJA.0000000000001059. PMID 31356373
- [Background] Dehghan F, Jalali R, Bashiri H. The effect of virtual reality technology on preoperative anxiety in children: a Solomon four-group randomized clinical trial. Perioper Med (Lond). 2019 Jun 4;8:5. doi: 10.1186/s13741-019-0116-0. eCollection 2019. PMID 31171963
- [Background] Jung MJ, Libaw JS, Ma K, Whitlock EL, Feiner JR, Sinskey JL. Pediatric Distraction on Induction of Anesthesia With Virtual Reality and Perioperative Anxiolysis: A Randomized Controlled Trial. Anesth Analg. 2021 Mar 1;132(3):798-806. doi: 10.1213/ANE.0000000000005004. PMID 32618627
- [Background] Ryu JH, Oh AY, Yoo HJ, Kim JH, Park JW, Han SH. The effect of an immersive virtual reality tour of the operating theater on emergence delirium in children undergoing general anesthesia: A randomized controlled trial. Paediatr Anaesth. 2019 Jan;29(1):98-105. doi: 10.1111/pan.13535. Epub 2018 Nov 25. PMID 30365231
- [Background] Ryu JH, Park SJ, Park JW, Kim JW, Yoo HJ, Kim TW, Hong JS, Han SH. Randomized clinical trial of immersive virtual reality tour of the operating theatre in children before anaesthesia. Br J Surg. 2017 Nov;104(12):1628-1633. doi: 10.1002/bjs.10684. Epub 2017 Oct 4. PMID 28975600
- [Background] Koo CH, Park JW, Ryu JH, Han SH. The Effect of Virtual Reality on Preoperative Anxiety: A Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Sep 29;9(10):3151. doi: 10.3390/jcm9103151. PMID 33003411
- [Background] Pasin L, Febres D, Testa V, Frati E, Borghi G, Landoni G, Zangrillo A. Dexmedetomidine vs midazolam as preanesthetic medication in children: a meta-analysis of randomized controlled trials. Paediatr Anaesth. 2015 May;25(5):468-76. doi: 10.1111/pan.12587. Epub 2015 Jan 6. PMID 25559766
- [Background] Fortier MA, Kain ZN. Treating perioperative anxiety and pain in children: a tailored and innovative approach. Paediatr Anaesth. 2015 Jan;25(1):27-35. doi: 10.1111/pan.12546. Epub 2014 Sep 30. PMID 25266082
- [Background] Agbayani CG, Fortier MA, Kain ZN. Non-pharmacological methods of reducing perioperative anxiety in children. BJA Educ. 2020 Dec;20(12):424-430. doi: 10.1016/j.bjae.2020.08.003. Epub 2020 Oct 21. No abstract available. PMID 33456927
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment took place during pre-anaesthetic assessment at the Hong Kong Children's Hospital pre-anaesthetic clinic between November 2022 to June 2024. The first patient was enrolled on 17 November 2022 and the last patient was enrolled on 5 June 2024. Of 114 participants enrolled, 84 met criteria and were randomized to treatment. The first patient assessment was on 3 January 2023. The last patient completed assessment 11 September 2024.
Pre-assignment Details: After patient enrollment, 30 of them dropped out before randomization due to surgery cancellation (n=10) , change of surgical plan (n=12), advancement or delay of surgery date resulting in children either too young or too mature for inclusion (n=4), or unavailability of researchers on surgery date (n=4).
Period: Overall Study
Arm/Group | Virtual reality (VR) group | Control group
Started | 42 | 42
Completed | 34 | 38
Not Completed | 8 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Incomplete data entry | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual reality (VR) group | Control group | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 38 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.94 (2.26) | 8.34 (2.02) | 8.16 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 24 | 34 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Surgery [Count of Participants; unit: Participants]
  General Surgery | 25 | 30 | 55
  Urology | 2 | 2 | 4
  Endocrine | 0 | 1 | 1
  Orthopaedics | 1 | 0 | 1
  Dental | 5 | 2 | 7
  Ear Nose Throat | 1 | 3 | 4
American Society of Anaesthesiologists (ASA) Physical Status Classification [Count of Participants; unit: Participants] — American Society of Anaesthesiologists (ASA) Physical Status Classification System, with classification as follows:
  ASA I = A normal healthy patient ASA II= A patient with mild systemic disease ASA III = A patient with severe systemic disease ASA IV = A patient with severe systemic disease that is a constant threat to life ASA V = A morbund patient who is not expected to survive with the operation ASA VI = A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA I | 30 | 30 | 60
    ASA II | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Modified Yale Preoperative Anxiety Scale (mYPAS) (T1)
Description: Primary outcome is whether there is a significant reduction of anxiety of children at induction, defined by a 20% change in the modified Yale Preoperative Anxiety Scale (mYPAS) between control group and intervention group at anaesthesia induction T1.
  mYPAS is considered the gold standard in assessing preoperative anxiety in children , consisting of 27 items divided into five domains: activity, emotional expressivity, state of arousal, vocalization and use of parents/legal guardians. The score ranges from minimum 23.3 to 100. A cut-off of >/= 30 indicates a high anxiety level in children. Higher score indicates increasing preoperative anxiety.
  This instrument has been considered as a gold standard instrument for measuring preoperative anxiety and had been administered in many previous studies. mYPAS will be assessed by a blinded researcher or anaesthesiologist, at induction in the operating theatre
Time Frame: During anaesthesia induction, from entering the operating theatre to successful anaesthesia induction (entered into state of general anaesthesia), usual time frame about 10 to 15 minutes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 34 | 38
score on a scale | 31.4 (8.2) | 37.3 (14.5)

2. Secondary Outcome: Baseline Preoperative Anxiety Score Using mYPAS on Admission (T0)
Description: After admission on the day of surgery, mYPAS assessment to be conducted preoperatively before randomization by a blinded researcher. mYPAS score (as stated in primary outcome measure description above) ranges from minimum 23.3 to 100. A cut-off of >/= 30 indicates a high anxiety level in children. Higher score indicates increasing preoperative anxiety.
Time Frame: Preoperative (at ward admission on day of surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 34 | 38
score on a scale | 34.8 (13.2) | 36.3 (17.3)

3. Secondary Outcome: Induction Compliance Checklist
Description: Score of checklist previously quoted in other literature that measures behaviours during anaesthesia induction, assessed by blinded observer. Items include crying, turning head away from mask, verbal refusal, verbalization of fear or worry, pushes mask away with hands/pushes nurse away, covers mouth/nose, hysterical crying, kicking/arching back, requires physical restraint, complete passivity. Score range from 0 to 10. Total maximum score is 10. High score indicates reduction in compliance to anaesthesia induction procedures.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 34 | 38
score on a scale | 0.824 (1.03) | 1.13 (1.55)

4. Secondary Outcome: Procedure Behaviour Rating Scale PBRS
Description: Observational tool developed by Melamed and colleagues (specifically Barbara G. Melamed and her team) in the 1970s-1980s as part of research on behavioral distress during medical procedures, particularly in pediatric populations. It is used to assess a patient's behavior during medical or dental procedures, particularly in contexts where anxiety, distress, or uncooperative behavior may arise.
  Domains Assessed:
  Common behaviors rated include:
  * Verbal resistance (crying, complaining).
  * Physical resistance (pulling away, flailing).
  * Facial expressions (grimacing, clenched teeth).
  * Cooperation level (following instructions, remaining still).
  Scoring:
  * Typically uses a Likert scale (e.g., 1-5) or categorical ratings (e.g., "none," "mild," "severe").
  * Higher scores indicate greater distress or noncompliance.
  * Maximum total score = 25 (Score range 0-25)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 34 | 38
score on a scale | 1.56 (1.76) | 1.92 (2.08)

5. Secondary Outcome: Parental Anxiety by State-trait Anxiety Inventory (STAI)-T
Description: Validated psychological assessment tool designed to measure anxiety in adults. Developed by Charles Spielberger, Richard Gorsuch, and Robert Lushene in 1970, it distinguishes between two types of anxiety:
  Trait Anxiety (STAI-T) measures a person's general tendency toward anxiety (how a person typically feels).
  STAI Including 40-item self-report questionnaire (20 items for state anxiety, 20 for trait anxiety).
  Scoring: Likert scale (1 to 4), with higher scores indicating higher anxiety levels.
  Total score ranged from 20-80 with higher score indicating more anxiety-prone personality (trait anxiety)
  Traditional Chinese validated version will be given to Chinese speaking parents.
Time Frame: during surgery, while parents waiting for children
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 34 | 38
score on a scale | 39 (10) | 41.8 (8.2)

6. Secondary Outcome: Parental Anxiety by State-trait Anxiety Inventory (STAI-S)
Description: Validated psychological assessment tool designed to measure anxiety in adults. Developed by Charles Spielberger, Richard Gorsuch, and Robert Lushene in 1970, it distinguishes between two types of anxiety:
  Validated psychological assessment tool designed to measure anxiety in adults. Developed by Charles Spielberger, Richard Gorsuch, and Robert Lushene in 1970, it distinguishes between two types of anxiety:
  State Anxiety (STAI-S) measures temporary, situational anxiety (how a person feels right now).
  STAI Including 40-item self-report questionnaire (20 items for state anxiety, 20 for trait anxiety).
  Scoring: Likert scale (1 to 4), with higher scores indicating higher anxiety levels.
  Score ranged from 20-80 with higher score indicating increasing current (state) anxiety.
  Traditional Chinese validated version will be given to Chinese speaking parents.
Time Frame: Parent to be completed in waiting room while waiting for participant to complete surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 34 | 38
score on a scale | 39.6 (11.1) | 43.3 (9.3)

7. Secondary Outcome: Parental Satisfactory Score
Description: Standard form to be given to every parent after general anaesthesia, with four-point scale (very unsatisfied(1), not satisfied(2), satisfied(3), very satisfied(4)) to 4 questions including
  * Are you satisfied with our preadmission service? (Pre-anaesthetic assessment/Pre-anaesthesia clinic)
  * Are you satisfied with our preoperative instructions?
  * Are you satisfied with the operating theatre service?
  * Are you satisfied with postoperative service? The total score is calculated as the sum of all items, range from minimum 4 to maximum 16. Higher score indicating higher satisfaction.
Time Frame: To be completed by parent after anaesthesia and to be submitted to research team on Day 1 post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual reality (VR) group | Control group
Number analyzed (Participants) | 32 | 34
score on a scale | 14.5 (1.8) | 14.0 (1.87)

ADVERSE EVENTS:
Time Frame: During implementation of virtual reality device on surgery day. The virtual reality device is given to child and monitored by Hospital Play Specialist and parent. The whole virtual reality experience lasted for approximately 10 to 15 minutes. Patient or parent may request to terminate the virtual reality experience at any time point during the application. Any adverse event happen during the application period will be recorded and collected.
Description: 1. All-cause mortality
  2. Serious Adverse Events: Discontinuation of virtual reality experience because of physical injury or discomfort (dizziness, nausea, vomiting, etc.) and that may require medical or surgical intervention
  3. Other (Not Including Serious) Adverse Events: Discontinuation of virtual reality experience because of physical discomfort that does not require medical or surgical intervention
Arm/Group | Virtual reality (VR) group | Control group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

LIMITATIONS AND CAVEATS:
1. Timing of VR exposure was standardized, and we did not evaluate whether the intervention's effectiveness differs when administered on the same day versus earlier before surgery.
2. Study focused primarily on anxiety reduction and induction compliance, without assessing other important aspects of the patient experience, such as pain perception, satisfaction, or overall healthcare experience from the child's perspective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT07018999/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT07018999/ICF_001.pdf